CLINICAL TRIAL: NCT02089919
Title: Study of Cancer Stem Cell Vcccinie That as a Specific Antigen in Metastatic Adenocarcinoma of the Liver
Brief Title: Cancer Stem Cells Vaccine Therapy in Treating Hepatocellular Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLH-001; 201401 (Other Grant/Funding Number: The research fund of Fuda cancer hospital in Guangzhou)
Record Dates: First submitted 2014-03-16; First posted 2014-03-18 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-03

CONDITIONS: Neoplasms, Liver
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- non-cancer stem cell vaccine (Placebo Comparator): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving low dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving middle dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine
- giving high dose vaccine (Experimental): The using dosage,frequency and duration of cancer stem cell vaccine are still undetermined.
  Interventions: Biological: cancer stem cell vaccine

INTERVENTIONS:
Biological: cancer stem cell vaccine

SUMMARY:
Most studies of cancer stem cells (CSC) involve the inoculation of cells from human tumors into immunosuppressed mice, preventing an assessment on the immunologic interactions and effects of CSCs. In this study, the investigators examined the vaccination effects produced by CSC-enriched populations from histologically distinct murine tumors after their inoculation into different syngeneic immunocompetent hosts. Enriched CSCs were immunogenic and more effective as an antigen source than unselected tumor cells in inducing protective antitumor immunity.Immune sera from CSC-vaccinated hosts contained high levels of IgG which bound to CSCs, resulting in CSC lysis in the presence of complement.CTLs generated from peripheral blood mononuclear cells or splenocytes harvested from CSC-vaccinated hosts were capable of killing CSCs in vitro. Mechanistic investigations established that CSC-primed antibodies and T cells were capable of selective targeting CSCs and conferring anti-tumor immunity.

DETAILED DESCRIPTION:
To assess the feasibility of generating CSC-loaded DC vaccines for clinical use, the investigators will harvest peripheral blood and tumor specimen from patients with hepatocellular cancer. The investigators will purify T, B cells and generate DCs from the PBMCs of the hepatocellular cancer patient.On the other hand, investigators will isolate ALDHhigh and ALDHlow tumor cells from the tumor specimen of the hepatocellular cancer patient using a similar protocol as investigators reported .

Aim 1: To demonstrate, in vitro, the relative cellular anti-hepatocellular cancer CSC immunity induced by hepatocellular cancer CSC-DC primed cytotoxic T cells.

Aim 2: To determine, in vitro, specific binding and lysis of hepatocellular cancer CSCs by antibodies produced by purified B cells from PBMCs stimulated with hepatocellular cancer CSC-DC.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients with a diagnosis of HCC based on histology or the current accepted radiological measures.
2. Age > 18 years.
3. Patient has an MRI or CT result (positive for HCC) up to 3 months prior to recruitment.
4. AFP >30.
5. Patient who is not eligible for or failed any HCC treatment.
6. Karnofsky performance status >70%.
7. The patient shows normal organ function according to the following parameters(as measured within six weeks prior to treatment allocation):

   Hemoglobin: Within normal range according to institutional standards; Absolute leukocyte count: Within normal range according to institutional standards; Absolute lymphocyte count: Within normal range according to institutional standards; Platelet count: Within normal range according to institutional standards; Alanine aminotransferase: ≤ 2.5 x Upper Limit of Normal (ULN); Aspartate aminotransferase: ≤ 2.5 x ULN; Total bilirubin: ≤ 1.5 x ULN. In the case of known Gilbert's syndrome ≤ 2 x ULN; Serum creatinine: 1.5 x ULN; Calculated creatinine clearance: > 50 mL/min .
8. No history of autoimmune diseases.
9. Ability to understand the study protocol and a willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients receiving anticoagulation therapy.
2. Patients who have received prior gemcitabine or radiation therapy to the liver bed.
3. Patients receiving any other investigational agents.
4. Patients with known brain metastases will be excluded because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse effects.
5. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
6. Patients who test positive for Hepatitis B virus, Hepatitis C virus or HIV. 7. level 3 hypertension; 8. severe coronary disease; 9. myelosuppression; 10. respiratory disease; 11. brain metastasis; 12. chronic infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The number of participants with adverse events | up to 3 months

SECONDARY OUTCOMES:
The secondary objectives are to evaluate vaccine immune responses to the immunizations by the data of body measurements | 1 month

OTHER OUTCOMES:
The dose of CSC vaccine | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Ning N, Pan Q, Zheng F, Teitz-Tennenbaum S, Egenti M, Yet J, Li M, Ginestier C, Wicha MS, Moyer JS, Prince ME, Xu Y, Zhang XL, Huang S, Chang AE, Li Q. Cancer stem cell vaccination confers significant antitumor immunity. Cancer Res. 2012 Apr 1;72(7):1853-64. doi: 10.1158/0008-5472.CAN-11-1400. PMID 22473314
- See also: Related Info — http://www.fudahospital.com/